CLINICAL TRIAL: NCT06183047
Title: Predictive Value of Early Changes of Chromogranin A Levels in Patients With Neuroendocrine Tumours Treated With PRRT
Status: Completed | Type: Observational
Sponsor: Military Institute od Medicine National Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: CgA dynamics
Record Dates: First submitted 2023-12-13; First posted 2023-12-27 (Actual); Last update posted 2023-12-27 (Actual); Status verified 2023-12

CONDITIONS: Early Release of Chromogranin A (CgA)
MeSH Terms: interventions — Genes, fms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 80 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patients with neuroendocrine tumours: We aimed to assess the predictive value of early release of chromogranin A (CgA) in patients with neuroendocrine tumours (NET) treated with peptide receptor radionuclide therapy (PRRT).
  Interventions: Diagnostic Test: early release of chromogranin A (CgA) in patients with neuroendocrine tumours (NET) treated with peptide receptor radionuclide therapy (PRRT).

INTERVENTIONS:
Diagnostic Test: early release of chromogranin A (CgA) in patients with neuroendocrine tumours (NET) treated with peptide receptor radionuclide therapy (PRRT). — early release of chromogranin A (CgA) in patients with neuroendocrine tumours (NET) treated with peptide receptor radionuclide therapy (PRRT).

SUMMARY:
The results of the study suggest that an early change in CgA levels might serve as a prognostic factor in NET patients treated with PRRT.

ELIGIBILITY:
Inclusion Criteria:

* confirmed NET
* peptide receptor radionuclide therapy (PRRT)

Exclusion Criteria:

* lack of patient consent to a clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with neuroendocrine tumours (NET) treated with peptide receptor radionuclide therapy (PRRT).
Sampling Method: Probability Sample
Enrollment: 38 (Actual)
Dates: Start 2016-10-01 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2023-09-30 (Actual)

PRIMARY OUTCOMES:
The CgA level change | 2016-2023
  We aimed to assess the predictive value of early release of chromogranin A (CgA) in patients with neuroendocrine tumours (NET) treated with peptide receptor radionuclide therapy (PRRT).

CONTACTS AND LOCATIONS:
Overall Officials: Andrzej Mazurek, MD, Principal Investigator — Military Institute of Medicine

IPD SHARING:
Plan to Share IPD: No